CLINICAL TRIAL: NCT01148147
Title: Prevention of Cardiac and Vascular Periprocedural Complications in Patients Undergoing Coronary Angiography or Angioplasty: Intracoronary Adenosine Administration to Prevent Periprocedural Myonecrosis in Elective Coronary Angioplasty. A Prospective Double-blind Randomized Trial.
Brief Title: Intracoronary Adenosine Administration to Prevent Periprocedural Myonecrosis in Elective Coronary Angioplasty
Acronym: PREVENT-ICARUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Giuseppe De Luca, MD, PhD, AOU Maggiore della Carita - Eastern Piedmont University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CE 93/09; 2009-013681-92 (Registry Identifier: EUDRACT)
Record Dates: First submitted 2010-06-07; First posted 2010-06-22 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2010-09

CONDITIONS: Coronary Angioplasty
Keywords: Adenosine; randomized trial; periprocedural myocardial necrosis; elective coronary angioplasty
MeSH Terms: interventions — Adenosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Intracoronary Placebo administration
  Interventions: Drug: Placebo
- Adenosine (Active Comparator): Intracoronary adenosine administration
  Interventions: Drug: Adenosine

INTERVENTIONS:
Drug: Adenosine — Intracoronary adenosine administration (180 ug for LCA and 120 ug for RCA)
  Arms: Adenosine
Drug: Placebo — Intracoronary Placebo administration
  Arms: Placebo

SUMMARY:
Aim of the study is to evaluate the benefits from adjunctive intracoronary administration of adenosin in elective patients undergoing coronary angioplasty.

DETAILED DESCRIPTION:
This study will investigate the effects of adjunctive intracoronary administration of adenosine on periprocedural myocardial infarction as compared to placebo.

This is a double-blind randomized trial single-center study. The enrollment will last 10 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective coronary angioplasty

Exclusion Criteria:

Marked Bradycardia (< 40 bpm)

* Previous allergy to adenosine
* Inability to sign the informed consent
* Asthma
* Elevated cardiac enzymes (troponin I o CK-MB)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Increase in troponin I (> 3 times the upper normal limit) | At 12 hours after the procedure

SECONDARY OUTCOMES:
MACE(death, MI, urgent target-vessel revascularization) | 72 hours
Angiographic Coronary flow, as evaluated by corrected TIMI frame count. | 1 minute after the final stent implantation

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe De Luca, MD, Principal Investigator — AOU Maggiore della Carità
Locations (1):
- Giuseppe De Luca, Novara, Italy

REFERENCES:
- [Derived] De Luca G, Iorio S, Venegoni L, Marino P. Evaluation of intracoronary adenosine to prevent periprocedural myonecrosis in elective percutaneous coronary intervention (from the PREVENT-ICARUS Trial). Am J Cardiol. 2012 Jan 15;109(2):202-7. doi: 10.1016/j.amjcard.2011.08.027. Epub 2011 Oct 14. PMID 22000773